CLINICAL TRIAL: NCT03490851
Title: The Effect of a Breakfast Meal Containing Oat β-glucan on Food Intake at a Subsequent Meal in Normal-weight and Overweight Subjects: A Randomized, Placebo-controlled Cross-over Study
Brief Title: The Effect of a Breakfast Meal Containing Oat β-glucan on Food Intake at a Subsequent Meal in Normal-weight and Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PEP-1613
Record Dates: First submitted 2018-03-26; First posted 2018-04-06 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Satiety

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oatmeal + OatWell28XF Intervention 1 (Experimental): 2g β-glucan
  Interventions: Other: Oatmeal + OatWell28CF Int 1
- Oatmeal + OatWell28XF Intervention 2 (Experimental): 4g β-glucan
  Interventions: Other: Oatmeal + OatWell28CF Int 2
- Oatmeal + OatWell28XF Intervention 3 (Experimental): 4g β-glucan plus β-glucanase
  Interventions: Other: Oatmeal + OatWell28CF Int 3
- Cream of Rice (Placebo Comparator): 27 grams of cream of rice
  Interventions: Other: Cream of Rice

INTERVENTIONS:
Other: Oatmeal + OatWell28CF Int 1 — Intervention involves consumption of one cereal in the beginning of each visit of the crossover sequence.
  Arms: Oatmeal + OatWell28XF Intervention 1
Other: Oatmeal + OatWell28CF Int 2 — Intervention involves consumption of one cereal in the beginning of each visit of the crossover sequence.
  Arms: Oatmeal + OatWell28XF Intervention 2
Other: Oatmeal + OatWell28CF Int 3 — Intervention involves consumption of one cereal in the beginning of each visit of the crossover sequence.
  Arms: Oatmeal + OatWell28XF Intervention 3
Other: Cream of Rice — Intervention involves consumption of one cereal in the beginning of each visit of the crossover sequence.
  Arms: Cream of Rice

SUMMARY:
The objectives of this study are to determine, in normal-weight and overweight subjects the effect of: Primary: oatmeal containing 4 g oat β-glucan on food intake at a subsequent meal compared to Cream of Rice cereal. Secondary: (i) oatmeal containing 2 g oat β-glucan on food intake at a subsequent meal compared to Cream of Rice cereal; and (ii) oatmeal containing 2g, 4g and 4g low MW oat beta-glucan on subjective appetite ratings, gastric emptying, postprandial responses of glucose, insulin, ghrelin and PYY levels compared to those elicited by Cream of Rice cereal. In addition, the relationship between amount, MW and viscosity of OBG and the primary and secondary objectives will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male or non-pregnant, non-lactating females, 18-60 years of age, inclusive.
* Subject is not currently participating nor recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement or lifestyle modification. Subject has not participated in another trial involving measurement of postprandial glucose response within 5 days of any of the 4 test visits in this study.
* Body mass index (BMI) ≥ 20.0 and < 30.0 kg/m² at screening.
* Unrestrained eater (<11)
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
* Willing to abstain from strenuous exercise, consuming alcoholic drinks 24 hours before study days and during study days.
* Willing to maintain current dietary supplement use throughout the trial. On test days, subject agrees not to take any dietary supplements until dismissal from the GI labs. Failure to comply will result in a rescheduled test visit.
* Normal fasting serum glucose (<7.0mmol/L capillary corresponding to whole blood glucose <6.3mmol/L).
* Hemoglobin ≥120g/L for females or ≥130g/L for males.
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria.
* Smokers
* Hemoglobin measurements of <120g/L for females and <130g/L for males (as per WHO criteria for anemia)
* Known history of AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders.
* Use of medications known to influence carbohydrate metabolism, gastrointestinal function or appetite, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or with any condition which might, in the opinion of Dr. Wolever, the president of GI Testing, either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Major trauma or surgical event within 3 months of screening.
* Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
* Known intolerance, sensitivity or allergy to any ingredients in the study test meals.
* Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.).
* Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg as defined by the average blood pressure measured at screening.
* Change in body weight of >3.5kg within 4 weeks of the screening visit.
* Presence of any signs or symptoms of an active infection within 5 d prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved and any treatment (i.e. antibiotic therapy) has been completed at least 5 d prior to each test visit.
* History of cancer in the prior two years, except for non-melanoma skin cancer.
* Recent history (within 12 months of screening) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as > 14 drinks per week (1 drink=12 oz beer, 5 oz wine, or 1.5 oz distilled spirits).
* Pregnancy or breastfeeding (pregnancy diagnosed on medical history at each visit)
* Any history of an eating disorder (e.g. anorexia nervosa, bulimia nervosa, binge eating) diagnosed by a qualified health professional.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-05-07 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Amount in caloric content of ingested food at a subsequent meal | 3 hours post consumption
  Amount in caloric content of ingested food at a subsequent meal in response to Oatmeal containing 4 g oat β-glucan compared to Cream of Rice cereal, in normal-weight and overweight subjects.

SECONDARY OUTCOMES:
Amount in caloric content of ingested food at a subsequent meal | 0-3 hours post consumption
  Amount in caloric content of ingested food at a subsequent meal in response to Oatmeal containing 2 g oat β-glucan compared to Cream of Rice cereal, in normal-weight and overweight subjects.
rate of gastric emptying | 0-3 hours post consumption
  after intake of oatmeal containing either 2g, 4g or 4g low MW oat beta-glucan
postprandial responses of blood glucose | 0-3 hours post consumption
  after intake of oatmeal containing either 2g, 4g or 4g low MW oat beta-glucan
postprandial responses of serum insulin | 0-3 hours post consumption
  after intake of oatmeal containing either 2g, 4g or 4g low MW oat beta-glucan
postprandial responses of gut hormone ghrelin | 0-3 hours post consumption
  after intake of oatmeal containing either 2g, 4g or 4g low MW oat beta-glucan
postprandial responses of gut hormone PYY | 0-3 hours post consumption
  after intake of oatmeal containing either 2g, 4g or 4g low MW oat beta-glucan
subjective ratings of appetite | 0-4.5 hours post consumption
  after intake of oatmeal containing either 2g, 4g or 4g low MW oat beta-glucan

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, MD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data
Time Frame: Late 2019

REFERENCES:
- [Derived] Wolever TMS, Tosh SM, Spruill SE, Jenkins AL, Ezatagha A, Duss R, Johnson J, Chu Y, Steinert RE. Increasing oat beta-glucan viscosity in a breakfast meal slows gastric emptying and reduces glycemic and insulinemic responses but has no effect on appetite, food intake, or plasma ghrelin and PYY responses in healthy humans: a randomized, placebo-controlled, crossover trial. Am J Clin Nutr. 2020 Feb 1;111(2):319-328. doi: 10.1093/ajcn/nqz285. PMID 31828287